CLINICAL TRIAL: NCT03119649
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled Study to Evaluate Multiple Doses of GLPG2222 in Subjects With Cystic Fibrosis Who Are Homozygous for the F508del Mutation
Brief Title: A Study to Evaluate Multiple Doses of GLPG2222 in Adult Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG2222-CL-202
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — GLPG2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A: GLPG2222 50 mg once daily (QD) (Experimental): Participants received a single GLPG2222 50 mg tablet and two matching placebo tablets orally, QD for 29 days.
  Interventions: Drug: GLPG2222 50 mg; Drug: Placebo
- Cohort A: GLPG2222 100 mg QD (Experimental): Participants received a single GLPG2222 100 mg tablet and two matching placebo tablets orally, QD for 29 days.
  Interventions: Drug: GLPG2222 100 mg; Drug: Placebo
- Cohort B: GLPG2222 200 mg QD (Experimental): Participants received two GLPG2222 100 mg tablets and one matching placebo tablet orally, QD for 29 days.
  Interventions: Drug: Placebo; Drug: GLPG2222 200 mg
- Cohort B: GLPG2222 400 mg QD (Experimental): Participants received two GLPG2222 150 mg tablets and one GLPG2222 100 mg tablet orally, QD for 29 days.
  Interventions: Drug: Placebo; Drug: GLPG2222 400 mg
- Cohort A Placebo (Placebo Comparator): Participants received three matching placebo tablets, orally, QD for 29 days.
  Interventions: Drug: Placebo
- Cohort B Placebo (Placebo Comparator): Participants received three matching placebo tablets, orally, QD for 29 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG2222 50 mg — Oral tablet(s) containing GLPG2222
  Arms: Cohort A: GLPG2222 50 mg once daily (QD)
Drug: GLPG2222 100 mg — Oral tablet(s) containing GLPG2222
  Arms: Cohort A: GLPG2222 100 mg QD
Drug: Placebo — Matching oral tablet(s) containing placebo
Drug: GLPG2222 200 mg — Oral tablet(s) containing GLPG2222
  Arms: Cohort B: GLPG2222 200 mg QD
Drug: GLPG2222 400 mg — Oral tablet(s) containing GLPG2222
  Arms: Cohort B: GLPG2222 400 mg QD

SUMMARY:
This is a Phase IIa, multi-center, randomized, double-blind, placebo-controlled, parallel-group study to evaluate 4 different doses of GLPG2222 administered for 4 weeks to adult subjects with a confirmed diagnosis of CF and homozygous for the F508del Cystic Fibrosis Transmembrane conductance Regulator (CFTR) mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥ 18 years of age, on the day of signing the Informed Consent Form (ICF).
2. A confirmed clinical diagnosis of CF and homozygous for the F508del CFTR mutation
3. Weight ≥ 40 kg.
4. Stable concomitant treatment for at least 4 weeks (28 days) prior to baseline
5. Forced expiratory volume in 1 second (FEV1) ≥ 40% of predicted normal for age, gender and height at screening

Exclusion Criteria:

1. History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
2. Unstable pulmonary status or respiratory tract infection requiring a change in therapy within 4 weeks of baseline.
3. Need for supplemental oxygen during the day, and >2 liters per minute (LPM) while sleeping.
4. Use of CFTR modulator therapy (e.g. lumacaftor or ivacaftor) within 4 weeks prior to the first study drug administration.
5. History of hepatic cirrhosis with portal hypertension.
6. Abnormal liver function test at screening; defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/ or alkaline phosphatase and/or gamma-glutamyl transferase (GGT) ≥ 3x the upper limit of normal (ULN); and/or total bilirubin (>1.5 times ULN)
7. Estimated creatinine clearance < 60 mL/min using the Cockcroft-Gault formula at screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van Steen, MD, MBA, Study Director — Galapagos NV
Locations (23):
- United States (7):
  - Child Health Research Unit at UAB, Chatom, Alabama
  - University of Arkansas for medical Sciences, Little Rock, Arkansas
  - Central Florida Pulmonary Group, Orlando, Florida
  - Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - Maine Medical Center, Portland, Maine
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina
- Belgium (4):
  - UZ Antwerpen, Antwerp
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Netherlands (4):
  - AMC Amsterdam, Amsterdam
  - Erasmus medisch centrum, Rotterdam
  - Haga Ziekenhuis, The Hague
  - UMC Utrecht, Utrecht
- Mother and child health institute of Serbia, New Belgrade, Serbia
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitarii Plitecnic La Fe, Valencia
- United Kingdom (4):
  - Papworth Hospital, Cambridge
  - St James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Southampton general Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bell SC, Barry PJ, De Boeck K, Drevinek P, Elborn JS, Plant BJ, Minic P, Van Braeckel E, Verhulst S, Muller K, Kanters D, Bellaire S, de Kock H, Geller DE, Conrath K, Van de Steen O, van der Ent K. CFTR activity is enhanced by the novel corrector GLPG2222, given with and without ivacaftor in two randomized trials. J Cyst Fibros. 2019 Sep;18(5):700-707. doi: 10.1016/j.jcf.2019.04.014. Epub 2019 May 3. PMID 31056441

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Participants received three matching placebo tablets orally, once a day (QD) for 29 days.
- Cohort A: GLPG2222 50 mg QD: Participants received a single GLPG2222 50 mg tablet and two matching placebo tablets, orally, QD for 29 days.
- Cohort A: GLPG2222 100 mg QD: Participants received a single GLPG2222 100 mg tablet and two matching placebo tablets, orally, QD for 29 days.
- Cohort B: GLPG2222 200 mg QD: Participants received two GLPG2222 100 mg tablets and one matching placebo tablet, orally, QD for 29 days.
- Cohort B: GLPG2222 400 mg QD: Participants received two GLPG2222 150 mg tablets and one GLPG2222 100 mg tablet, orally, QD for 29 days.
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Started | 11 | 10 | 10 | 14 | 14
Completed | 11 | 10 | 10 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least one dose of study drug.
Groups:
- Pooled Placebo: Participants received three matching placebo tablets orally, QD for 29 days.
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD | Total
Number analyzed (Participants) | 11 | 10 | 10 | 14 | 14 | 59
Age, Continuous [Median (Full Range); unit: years] | 27.0 [21 to 58] | 26.0 [20 to 37] | 24.0 [18 to 35] | 32.0 [19 to 47] | 26.0 [19 to 59] | 27.0 [18 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 7 | 5 | 25
  Male | 7 | 7 | 4 | 7 | 9 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unknown data were not reported because local regulations did not allow the Sponsor to ask for the information.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 11 | 9 | 10 | 13 | 13 | 56
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of participants with any treatment-emergent adverse events (TEAEs) and serious or treatment-related TEAEs, as well as number of patients with TEAEs by worst intensity reported (mild, moderate, or severe).
Time Frame: First administration (Day 1) through Follow-up (Day 43)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 11 | 10 | 10 | 14 | 14
Participants
  Any TEAE | 9 | 8 | 10 | 11 | 9
  Any Serious TEAE | 2 | 0 | 1 | 0 | 0
  Worst TEAE Intensity=Mild | 6 | 4 | 7 | 8 | 9
  Worst TEAE Intensity=Moderate | 2 | 4 | 2 | 2 | 0
  Worst TEAE Intensity=Severe | 1 | 0 | 1 | 1 | 0
  Any Treatment-related TEAE | 2 | 2 | 6 | 5 | 1

2. Secondary Outcome: Mean Change From Baseline in Sweat Chloride Concentration at Day 29
Description: Two sweat collections, one from each arm, were obtained. Mean sweat chloride concentration was determined from both arms and measured as millimoles per liter (mmol/L). Baseline was defined as the predose value on Day 1 (or the last non-missing predose measurement).
Time Frame: Prior to dosing on Days 1 and 29, or at early discontinuation
Population: Intent-to-treat (ITT) population: all enrolled participants who received at least one dose of study drug and had at least one post-baseline assessment with efficacy data. Only participants with non-missing data at baseline were included in the analysis; 3 participants had missing sweat chloride concentration data at baseline.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 11 | 9 | 8 | 14 | 14
mmol/L | -2.5 (2.79) | -5.8 (3.08) | -6.6 (3.29) | -18.3 (2.49) | -8.8 (2.49)
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: GLPG2222 50 mg QD; Day 29: GLPG2222 50 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.4291, ANCOVA — P-value obtained from the Mixed Effects Model for Repeated Measures (MMRM) analysis with treatment as factor and baseline as covariate. Pairwise comparisons were not corrected for multiplicity; Difference in LS Means = -3.3, 95% CI 2-sided [-11.6 to 5.0], Standard Error of Mean 4.15
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort A: GLPG2222 100 mg QD; Day 29: GLPG2222 100 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.3477, ANCOVA — P-value obtained from the MMRM analysis with treatment as factor and baseline as covariate. Pairwise comparisons were not corrected for multiplicity; Difference in LS Means = -4.10, 95% CI 2-sided [-12.8 to 4.6], Standard Error of Mean 4.32
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort B: GLPG2222 200 mg QD; Day 29: GLPG2222 200 mg QD vs. Pooled Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = -15.8, 95% CI 2-sided [-23.2 to -8.3], Standard Error of Mean 3.72
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: GLPG2222 400 mg QD; Day 29: GLPG2222 400 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.0995, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = -6.3, 95% CI 2-sided [-13.9 to 1.2], Standard Error of Mean 3.76

3. Secondary Outcome: Mean Change From Baseline in Percent (%) Predicted FEV1 (%FEV1) at Day 29
Description: Percent predicted FEV1 for age, gender, and height was determined from standardized spirometry assessments and estimated using the 2012 Global Lungs Initiative equation. Baseline was defined as the last non-missing predose assessment on Day 1.
Time Frame: Predose and between 1 and 2 hours postdose on Days 1 and 29, or at early discontinuation
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: % predicted FEV1
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 11 | 10 | 10 | 14 | 14
% predicted FEV1 | -1.0 (1.45) | 0.1 (1.50) | -0.3 (1.51) | 0.0 (1.27) | 1.3 (1.26)
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: GLPG2222 50 mg QD; Day 29: GLPG2222 50 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.5940, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 1.1, 95% CI 2-sided [-3.1 to 5.4], Standard Error of Mean 2.11
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort A: GLPG2222 100 mg QD; Day 29: GLPG2222 100 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.7553, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 0.6, 95% CI 2-sided [-3.5 to 4.8], Standard Error of Mean 2.06
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort B: GLPG2222 200 mg QD; Day 29: GLPG2222 200 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.5958, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 1.0, 95% CI 2-sided [-2.9 to 4.9], Standard Error of Mean 1.94
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: GLPG2222 400 mg QD; Day 29: GLPG2222 400 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.2403, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 2.3, 95% CI 2-sided [-1.6 to 6.2], Standard Error of Mean 1.94

4. Secondary Outcome: Mean Change From Baseline in the Respiratory Domain of the Cystic Fibrosis Questionnaire-Revised (CFQ-R) at Day 29
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. The respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), derived from Questions 40, 41, 42, 45, and 46 if at least 50% of the questions had non-missing data. The scale score ranged from 0-100; higher scores indicated fewer symptoms and better health-related quality of life with a negative change indicating a worsening of symptoms. A change of 4 is considered clinically relevant.
Time Frame: Prior to dosing on Days 1 and 29, or at early discontinuation
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 11 | 10 | 10 | 14 | 14
units on a scale | -2.4 (3.32) | 0.4 (3.47) | -0.7 (3.48) | 4.5 (2.93) | -0.8 (2.93)
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort A: GLPG2222 50 mg QD; Day 29: GLPG2222 50 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.5749, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 2.7, 95% CI 2-sided [-6.9 to 12.4], Standard Error of Mean 4.81
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort A: GLPG2222 100 mg QD; Day 29: GLPG2222 100 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.7381, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 1.6, 95% CI 2-sided [-8.1 to 11.3], Standard Error of Mean 4.83
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort B: GLPG2222 200 mg QD; Day 29: GLPG2222 200 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.1282, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 6.8, 95% CI 2-sided [-2.0 to 15.7], Standard Error of Mean 4.43
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: GLPG2222 400 mg QD; Day 29: GLPG2222 400 mg QD vs. Pooled Placebo; Test type: Superiority; p = 0.7212, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Difference in LS Means = 1.6, 95% CI 2-sided [-7.3 to 10.5], Standard Error of Mean 4.43

5. Secondary Outcome: Mean Maximum Observed Plasma Concentration (Cmax; Nanograms Per Milliliter [mg/mL]) of GLPG2222
Description: Maximum concentration of GLPG2222 after multiple dosing (ng/ML), obtained directly from the observed concentration versus time data. All pharmacokinetic (PK) parameters were determined from Day 15; Day 29 data were determined if the participant was not available for full PK profiling on Day 15.
Time Frame: Day 15 (predose and 0.5, 1, 2, 3, 4, 6, and 8 hours postdose) and prior to dosing on Day 29
Population: Pharmacokinetic (PK) Population: all participants who were exposed to GLPG2222 and who had available and evaluable PK data (excluding all protocol violations/deviations or adverse events that may have had an impact on the PK analysis). Data were not calculable for 1 patient.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 10 | 10 | 14 | 13
ng/mL | 478 (128) | 1170 (395) | 2490 (535) | 5330 (2700)

6. Secondary Outcome: Mean GLPG2222 Plasma Concentration Observed at Predose (Ctrough; ng/mL)
Description: Plasma concentration of GLPG2222 observed at pre-dose (ng/mL), obtained directly from the observed concentration versus time data. Ctrough was calculated using both Day 15 and Day 29 PK data.
Time Frame: Days 15 and 29 (predose)
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 10 | 10 | 14 | 14
ng/mL | 48.1 (33.7) | 132 (87.2) | 343 (204) | 677 (659)

7. Secondary Outcome: Median Time to Occurrence of GLPG2222 Cmax (Tmax; Hours [h])
Description: Time of occurrence of maximum concentration of GLPG2222 after multiple dosing (h), obtained directly from the observed concentration versus time data. All PK parameters were determined from Day 15; Day 29 data were determined if the participant was not available for full PK profiling on Day 15.
Time Frame: Day 15 (predose and 0.5, 1, 2, 3, 4, 6, and 8 hours postdose) and prior to dosing on Day 29
Population: PK Population; data were not calculable for 1 patient.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 10 | 10 | 14 | 13
hours | 2.0 [1.0 to 6.0] | 2.0 [2.0 to 6.0] | 3.0 [2.0 to 4.0] | 2.0 [0.5 to 6.0]

8. Secondary Outcome: Mean Area Under the Concentration-Time Curve From Time 0 up to 24 Hours Following Multiple Dosing (AUC[0-t]; ng.h/mL) of GLPG2222
Description: Area under the concentration-time curve from time 0 up to 24 hours following multiple dosing (ng.h/mL), calculated by linear up/log down trapezoidal summation. All PK parameters were determined from Day 15; Day 29 data were determined if the participant was not available for full PK profiling on Day 15.
Time Frame: Day 15 (predose and 0.5, 1, 2, 3, 4, 6, and 8 hours postdose) and prior to dosing on Day 29
Population: PK Population; data were not calculable for 1 patient.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
Number analyzed (Participants) | 10 | 10 | 14 | 13
ng.h/mL | 3850 (1670) | 9670 (3770) | 22900 (7530) | 46400 (25500)

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form (ICF; Screening, Day -28) until the final follow-up visit (Day 43)
Arm/Group | Pooled Placebo | Cohort A: GLPG2222 50 mg QD | Cohort A: GLPG2222 100 mg QD | Cohort B: GLPG2222 200 mg QD | Cohort B: GLPG2222 400 mg QD
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/10 | 1/10 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 9/11 | 8/10 | 10/10 | 11/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=11) | Cohort A: GLPG2222 50 mg QD (N=10) | Cohort A: GLPG2222 100 mg QD (N=10) | Cohort B: GLPG2222 200 mg QD (N=14) | Cohort B: GLPG2222 400 mg QD (N=14)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=11) | Cohort A: GLPG2222 50 mg QD (N=10) | Cohort A: GLPG2222 100 mg QD (N=10) | Cohort B: GLPG2222 200 mg QD (N=14) | Cohort B: GLPG2222 400 mg QD (N=14)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 3 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Decreased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory depth decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sputum decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 2 | 1 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 3 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 3 | 5 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Retrograde amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 1
Exercise tolerance increased (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0
Thrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Azoospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must agree that before publishing or communicating any results of the trial, the sponsor has at least 90 days for full review of the information prior to submission.

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03119649/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT03119649/SAP_001.pdf